CLINICAL TRIAL: NCT00921297
Title: Therapeutic Effects of Cataract Removal in Alzheimer's Disease
Brief Title: Cataract Removal and Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other); MetroHealth Medical Center (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Grover C. Gilmore, PhD., Principal Investigator, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 04-09-21; 1R01AG030114 (NIH)
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Cataracts; Alzheimer's Disease
Keywords: Alzheimer's Disease; vision impairment; cataract; quality of life; retinal nerve fiber layer
MeSH Terms: conditions — Cataract; Alzheimer Disease; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Cataract Surgery (Active Comparator): Subjects randomly selected into the Immediate Surgery group will have their cataract surgery scheduled one month from the time their initial study visits are completed. The subjects will be followed monthly for a period of 6 months for surgical and non-surgical adverse events. At the 6-month point, subjects will receive a final comprehensive eye exam and neuropsychological testing. The research partners will complete final activities of daily living and resource utilization questionnaires.
  Interventions: Procedure: Immediate Cataract Surgery
- Delayed Cataract Surgery (No Intervention): Subjects selected into the Delayed Surgery group will be asked to delay their surgery for 6 months after their initial study visits. At 6 months, this group will also undergo the same testing as the Surgery Group.

INTERVENTIONS:
Procedure: Immediate Cataract Surgery — Cataract surgery, as part of standard of care, will be performed on 1/2 of the group under investigation.
  Arms: Immediate Cataract Surgery

SUMMARY:
Two very common aging-related diseases in older adults are Alzheimer's disease (AD) and cataracts. In elderly adults, these two diseases frequently occur in the same person. Although a cure for AD is currently unavailable, cataracts can be effectively treated with surgery in most people. The removal of cataracts has documented benefits for visual performance and for reducing accidents and falls. However, it has been the experience of the ophthalmologists, and others in the field, that patients, caregivers, and primary care doctors are reluctant to proceed with cataract surgery once an individual is given the diagnosis of AD. It is thought that cataract surgery will not improve the AD patient's quality of life, vision, and cognition. The investigators have designed this study to determine whether or not this is true.

DETAILED DESCRIPTION:
In this project, we propose to test the following clinical hypothesis, while addressing the primary and two secondary Specific Aims:

Hypothesis: Cataract removal produces measurable benefits in vision, perception, independent function, and quality of life in patients with co-morbid Alzheimer's disease.

Primary Specific Aim: To determine the effects of cataract removal on visual acuity, spatial contrast sensitivity, vision dependent functions, visual information processing, and quality of life in patients with Alzheimer's disease.

Secondary Specific Aims.

1. To delineate the baseline characteristics of those patients who benefit most from the surgical intervention.
2. To assess the thickness of the retinal nerve fiber layer (RNFL) with optical coherence tomography (OCT) in large samples of AD patients classified with mild or moderate dementia to determine if the thickness of the RNFL is associated with dementia severity, visual performance measures, and other patient characteristics.

The study is designed as a Randomized Controlled Trial (RCT) with two cohorts of AD patients in a longitudinal investigation. Each person will be evaluated periodically over a 6 month period. All participants will be diagnosed with visually significant bilateral cataractous lens. The cohorts will be established by randomly assigning patients to either the immediate or the (optional) delayed surgery group. Patients will be stratified by AD severity (CDR mild or moderate) and cataract severity prior to being randomized. Comparisons between and within groups will test the change over time in vision, visual information processing, and quality of life associated with or without the removal of cataracts. The RNFL thickness of each person will be evaluated with optical coherence tomography (OCT). The thickness of the RNFL will be compared across dementia severity levels. Each consented participant will have a consenting study partner who may be referred to as a Research Partner, and who will often be the participant's caregiver. The latter will help to assure protocol adherence by the AD participants and will provide information about behavioral symptoms, activities of daily living, and amount of resources used. The study will demonstrate the clinical efficacy of cataract removal as a direct intervention to potentially improve the visual and cognitive functions, and the quality of life in persons diagnosed with AD.

ELIGIBILITY:
Inclusion Criteria:

* age 50 and older
* clinical diagnosis of possible/probable Alzheimer's disease, or other type of dementia, mild (CDR-1), moderate (CDR-2), or severe (CDR-3)
* at least 1 visually significant cataract
* no ocular pathology
* psychotropic drug must be with stable dosage for 30 days

Exclusion Criteria:

* history of cataract removal
* history of visually significant retinal, or optic nerve abnormalities
* informed consent cannot be obtained from either subject or their research partner
* subject shows evidence (in preoperative testing) of unstable cardiac or pulmonary function
* history of uncontrolled diabetes or hypertension
* history of stroke in areas known to affect cognition
* life expectancy of less than 1 year
* Down's Syndrome

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-06; Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Visual acuity, spatial contrast sensitivity, visual perception and cognition | Baseline and Month 6

SECONDARY OUTCOMES:
Independent function | Baseline and Month 6
Quality of Life | Baseline and Month 6
Retinal Nerve Fiber Layer | Baseline, Months 2,4, & 6

CONTACTS AND LOCATIONS:
Overall Officials: Grover C. Gilmore, PhD., Principal Investigator — Case Western Reserve University; Sara Debanne, PhD., Study Director — Case Western Reserve University; Julie Belkin, M.D., Study Director — University Hospitals Cleveland Medical Center; Jonathan Lass, M.D., Study Director — University Hospitals Cleveland Medical Center; Alan Lerner, M.D., Study Director — University Hospitals Cleveland Medical Center; Thomas Steinemann, M.D., Study Director — MetroHealth Medical Center
Locations (2):
- United States (2):
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio